CLINICAL TRIAL: NCT00642057
Title: Compassionate Use of Tetrabenazine in the Treatment of Hyperkinesias
Brief Title: Compassionate Use of Tetrabenazine in the Treatment of Abnormal Movements
Acronym: TBZ
Status: No longer available | Type: Expanded Access
Sponsor: Joseph Jankovic (Other)
Responsible Party: Sponsor-Investigator, Joseph Jankovic, Professor, Neurology-PDCMDC, Baylor College of Medicine
Organization: Baylor College of Medicine (Other)
Other Study IDs: H-721
Record Dates: First submitted 2007-12-28; First posted 2008-03-24 (Estimated); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Hyperkinetic Movement Disorders
Keywords: chorea; dyskinesia; hyperkinetic
MeSH Terms: conditions — Chorea; Dyskinesias | interventions — Tetrabenazine

INTERVENTIONS:
Drug: tetrabenazine — 25 mg titrated to optimal dose per patient

SUMMARY:
Although the results of studies looking at tetrabenazine have shown its effectiveness in the management of hyperkinetic(too much) movement disorders, it has not been made available in the U.S. The drug must be obtained from Cambridge Laboratories, the distributor, using an individual IND (#16,161). The cost of the drug is passed on to the patient. The purpose of the protocol is to provide an efficacious drug, with few side effects, in an attempt to get rid of a variety of incapacitating dyskinesias (abnormal movements).

DETAILED DESCRIPTION:
The purpose of the protocol is to provide compassionate use of an efficacious drug, with few side effects, in an attempt to get rid of a variety of incapacitating dyskinesias (abnormal movements).

ELIGIBILITY:
Inclusion Criteria:

* Subjects evaluated here at Baylor in the PDCMDC demonstrating need for tetrabenazine treatment.
* Willing to sign informed consent.
* Willing to comply with procedures required as part of this study.

Exclusion Criteria:

* Those subjects unwilling to comply with study requirements.
* Subjects unable to give informed consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

REFERENCES:
- See also: Parkinson's Disease Center and Movement Disorders Clinic — http://www.jankovic.org